CLINICAL TRIAL: NCT05198986
Title: Effects of Pronation on Respiratory System Mechanical Properties and Ventilation in Patients With Acute Respiratory Distress Syndrome During Vv-ecmo
Brief Title: Pronation During Veno-venous Extra Corporeal Membrane Oxygenation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Prof, University Magna Graecia
Other Study IDs: ECMO-PP
Record Dates: First submitted 2022-01-03; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Respiratory Failure
Keywords: Extra Corporeal Membrane Oxygenation; Prone Position
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECMO Prone Position: After baseline assessment in supine position, patients will be positioned in prone position to assess modification of lung mechanics, aeration and hemodynamics
  Interventions: Other: Prone Position during Extra Corporeal Membrane Oxygenation (ECMO)

INTERVENTIONS:
Other: Prone Position during Extra Corporeal Membrane Oxygenation (ECMO) — Pronation will be executed according to a predefined protocol: 4 caregivers will be required for the procedure, one of them being dedicated to the management of the head of the patient, the endotracheal tube and the ventilator lines. The others will stand at each side of the bed. In the first step, the direction of the rotation will be decided giving priority to the side of the central venous lines. The patient will be then moved along the horizontal plane to the opposite side of the bed selected for the direction of rotation. In the third step, the patient will be moved in the sagittal plane and maintained in that position for a short while to attach the cardiac electrodes to her/his back and to set a new bed sheet. In the last step, the patient will be turned to the complete prone position.

SUMMARY:
The Acute Respiratory Distress Syndrome (ARDS) is defined by a recent (within 1 week) respiratory failure, not fully explained by cardiac failure or fluid overload. ARDS is also characterized by bilateral opacities at the chest imaging, with an alteration of the oxygenation while positive end-expiratory pressure equal or greater than 5 cmH2O is applied. Severe ARDS is characterized by a high mortality. In the most severe ARDS patients, venovenous extracorporeal membrane oxygenation (vv-ECMO) is increasingly accepted as a mean to support vital function, although not free from complications.

In patients with severe ARDS, prone position has been used for many years to improve oxygenation. In these patients, early application of prolonged (16 hours) prone-positioning sessions significantly decreased 28-day and 90-day mortality. More recently, prone position and ECMO have been coupled as concurrent treatment. Indeed, the addition of prone positioning therapy concurrently with ECMO can aid in optimizing alveolar recruitment, and reducing ventilator-induced lung injury. Nowadays, few data exist on respiratory mechanics modifications before and after the application of prone position in patients with severe ARDS receiving vv-ECMO. The investigators have therefore designed this observational study to assess the modifications of mechanical properties of the respiratory system, ventilation and aeration distribution, and hemodynamics occurring during ECMO before and after prone position in patients with severe ARDS.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients with a diagnosis of severe Acute Respiratory Distress Syndrome receiving veno-venous ECMO

Exclusion Criteria:

* mechanical ventilation for 7 days or longer
* pregnancy
* body mass index (BMI) > 45 kg/m2
* chronic respiratory failure with long-term oxygen therapy or domiciliary non-invasive ventilation
* cardiac failure resulting in veno-arterial ECMO
* history of heparin- induced thrombocytopenia
* cancer with a life expectancy of less than 5 years
* moribund condition or a Simplified Acute Physiology Score (SAPS-II) value of more than 90;
* current non drug- induced coma after cardiac arrest or presence of an irreversible neurologic injury
* decision to withhold or withdraw life--sustaining therapies
* presence of pneumothorax and/or pulmonary emphysema
* recent (1 week) thoracic surgery
* presence of chest burns
* inclusion in other research protocols
* refusal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will receive deep sedation and continuous infusion of neuromuscular blocking agents. Protective mechanical ventilation will be set in volume-controlled mode.
  A pulmonary artery catheter (PAC) will be also positioned and connected to a dedicated system for hemodynamic monitoring.
  After enrolment, a silicon 16-electrode belt of proper size will be positioned around the patient's chest between the 4th and 6th intercostal spaces and connected to the EIT device. The position of EIT belt will be therefore marked on the skin with a dermographic pencil to avoid its displacement. Invasive mechanical ventilation will be applied with a ventilator connected to the EIT device through a RS232 interface.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Driving Pressure | 30 minutes after the prone positioning
  Difference between the airway plateau pressure and the total positive end-expiratory pressure after an inspiratory and expiratory hold maneuvers, respectively

SECONDARY OUTCOMES:
Respiratory system compliance | 30 minutes after the prone positioning
  Driving pressure to the tidal volume ratio
Cardiac output | 30 minutes after the prone positioning
  Liters of blood flow ejected from the heart per minute, measured through a pulmonary artery catheter
Pulmonary arterial pressure | 30 minutes after the prone positioning
  pulmonary arterial pressure measured through a pulmonary artery catheter
End-Expiratory Lung Impedance | 30 minutes after the prone positioning
  Measurement of the end expiratory lung volume, as assessed by the electrical impedance tomography

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna graecia University
Locations (1):
- Federico Longhini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
Deindividualized data will be share on reasonable request to the Principal Investigator after study completion and publication
Supporting Information: Study Protocol
Time Frame: Data will be available after study completion and publication
Access Criteria: On reasonable request